CLINICAL TRIAL: NCT02407548
Title: The Effects of Dietary Supplement of Coenzyme Q10 on Dyslipidemia
Brief Title: The Effects of Dietary Supplement of Coenzyme Q10（CoQ10） on Dyslipidemia
Acronym: TEDSCD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, zhangpeiwen, PhD candidate, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SunYat-senU002
Record Dates: First submitted 2015-03-25; First posted 2015-04-03 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Dyslipidemia
Keywords: cholesterol efflux; dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- combined group (Experimental): each coenzyme Q10 vitamin E softgel contain CoQ 10 30mg + vitamin E 16mg; The subjects in this arm take 2 softgels after lunch and supper respectively per day. Total supplementation is 120mgCoQ10 and 64mg vitamin per day. The duration is 24 weeks.
  Interventions: Dietary Supplement: coenzyme Q10 vitamin E softgel
- CoQ10 group (Experimental): each softgel contain CoQ 10 30mg; The subjects in this arm take 2 softgels after lunch and supper respectively per day. Total supplementation is 120mgCoQ10 per day. The duration is 24 weeks.
  Interventions: Dietary Supplement: coenzyme Q10 softgel
- placebo group (Other): each softgel contain no vitamin E, no CoQ10; The subjects in this arm take 2 softgels after lunch and supper respectively per day. The duration is 24 weeks.
  Interventions: Dietary Supplement: placebo softgel

INTERVENTIONS:
Dietary Supplement: coenzyme Q10 vitamin E softgel — 4 coenzyme Q10 and vitamin E softgels per day for 24 weeks. Keep normal lift style unchanged.
  Arms: combined group
Dietary Supplement: coenzyme Q10 softgel — 4 coenzyme Q10 softgels per day for 24 weeks. Keep normal lift style unchanged.
  Arms: CoQ10 group
Dietary Supplement: placebo softgel — 4 placebo softgels per day. Keep normal lift style unchanged.
  Arms: placebo group

SUMMARY:
In previous study the investigators found that CoQ10 can improve cholesterol efflux from macrophages in cell model, ApoE mice model and small-scale of healthy volunteers. In addition, CoQ10 has strong antioxidant activity and is an essential factor of mitochondria electron transport chain. So the investigators hypothesize that CoQ10 may have some health promotion effect on dyslipidemia, risk factor of atherosclerosis and other cardiovascular diseases. On this purpose, the investigators are going to recruit 150 dyslipidemia patients to supply CoQ10+vitamin E or CoQ10 alone or placebo in different doses for 24 weeks to explore the effects of CoQ10 on cholesterol efflux and lipid profiles on dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* The subjects were considered to have dyslipidemia if they met 2 of the following 4 criteria:

  * fasting total cholesterol concentration>200 mg/dL,
  * fasting triglyceride concentration>150mg/dL,
  * fasting LDL-cholesterol concentrations>100 mg/dL, or
  * fasting HDL-cholesterol concentrations>40 mg/dL.

Exclusion Criteria:

* history of CVD or other severe chronic disease or use of any drugs known to affect lipid metabolism.
* use any antioxidant such as Vitamin E, vitamin C,Phytochemicals and coenzyme Q10 within two months before trial.
* pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Effects of CoQ10 on lipid profile | 6 months
  Tg, Tc, LDL, HDL, APOA1,APOB

SECONDARY OUTCOMES:
Effects of CoQ10 on blood glucose and insulin | 6 mouth
  reflect insulin sensibility
Effects of CoQ10 on oxidative stress and inflammation | 6 mouth

OTHER OUTCOMES:
Effects of CoQ10 on FGF21 | 6 month
  reflect glucose and lipid metabolism
Effects of CoQ10 on cholesterol efflux from macrophages | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: ling wenhua, professor, Study Director — SUN YAY-SEN UNIVERSITY
Locations (1):
- Hongshan Street community health service centre, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang P, Chen K, He T, Guo H, Chen X. Coenzyme Q10 supplementation improves adipokine profile in dyslipidemic individuals: a randomized controlled trial. Nutr Metab (Lond). 2022 Mar 3;19(1):13. doi: 10.1186/s12986-022-00649-5. PMID 35241098
- [Derived] Zhang P, Yang C, Guo H, Wang J, Lin S, Li H, Yang Y, Ling W. Treatment of coenzyme Q10 for 24 weeks improves lipid and glycemic profile in dyslipidemic individuals. J Clin Lipidol. 2018 Mar-Apr;12(2):417-427.e5. doi: 10.1016/j.jacl.2017.12.006. Epub 2017 Dec 21. PMID 29454678